CLINICAL TRIAL: NCT03678402
Title: Testing the Effectiveness of a Falls Prevention System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tammy Moore (Other)
Responsible Party: Sponsor-Investigator, Tammy Moore, Director of Nursing, Neurological Institute, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018H0303
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Results first posted 2022-01-04 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: High Risk for Falling
Keywords: falling; inpatient
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: single arm prospective non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Palarum Fall Prevention System (Experimental): The Study site, the OSU Wexner Center Brain and Spine Hospital, is located on three contiguous floors with each floor being made up of two units or Pods designated East and South. Following commencement of the study, and throughout its duration, Pods assigned to the Study will only utilize the Palarum Fall Prevention System and a monitored PUP™ sock, i.e., (Patient is Up) System as the standard of care intervention for fall prevention in accordance with its operating instructions and procedures.
  Interventions: Device: PUP™ sock

INTERVENTIONS:
Device: PUP™ sock — The Palarum Fall Prevention System that includes the PUP™ (Patient is Up) System, is made upon of seven tangible elements: an inpatient room Android tablet (IRT), a nurse station Android monitor (HUC), a local server (PLS), a cloud server (PCS), a Bluetooth Low Energy beacon(s), an Android smart watch, and an e-textile sock connected sensor transmitter (PUP™ sock). The PUP™ sock monitors and transmits pressure, force, acceleration and motion data.
  Other Names: PUP™ (Patient is Up) System

SUMMARY:
The purpose of this single arm intervention study is to determine if the fall rate (as measured by falls per 1000 patient days) for patients designated "high fall risk" decreases with the use of the PUP™ [Patient is UP Falls Prevention System] when compared to the historical falls rate data for the prior 12 months from those same nursing units within the OSUWM Brain & Spine Hospital.

DETAILED DESCRIPTION:
The purpose of this single arm intervention study is to determine if the fall rate (as measured by falls per 1000 patient days) for patients designated "high fall risk" decreases with the use of the PUP™ [Patient is UP Falls Prevention System] when compared to the historical falls rate data for the prior 12 months from those same nursing units within the OSUWM Brain & Spine Hospital. All Brain and Spine Hospital patients will be evaluated as to fall risk using the current fall risk assessment tool employed by OSU Medical Center and administered in the usual and customary fashion upon evaluation on the floor and Pod. Patients who are determined to be at a high fall risk will be approached to participate. Those patients who consent to participate in the study will remain in the study until a nurse removes the patient from high risk fall status or the participant has been discharged from the hospital. Any patient fall will to be reported and evaluated following current processes and procedures developed by the OSU Brain and Spine Institute as maintained with IHIS; the PUP™ as the intervention for this study will be an adjunct to those fall prevention processes already in place.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older;
* All high-risk fall patients, eighteen years of age or older, who are admitted to the OSU Brain and Spine Hospital on Floors 8 South, 9 South, 10 South, 8 East, 9 East or 10 East. Patients will undergo a pre-assessment as per OSUWMC procedure to determine if they are a high-fall risk.

Exclusion Criteria:

* Patients whose medical condition as assessed by the PI prohibits their participation in the program, which would include among others the following: patients who lack the capacity to consent, patients with an anatomy or wound issue on their feet or around their calves that would bar them from wearing socks on either foot, and/or patients for whom the sock would impede medical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Moore, RN, PHD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the institution. Any data to be shared will have been deidentified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palarum Fall Prevention System
Started | 521
Completed | 521
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Palarum Fall Prevention System
Number analyzed (Participants) | 521
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 425
  >=65 years | 96
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [18.1 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Was not reported in the study
  Male | NA — Was not reported in the study
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Not collected
  Asian | NA — Not collected
  Native Hawaiian or Other Pacific Islander | NA — Not collected
  Black or African American | NA — Not collected
  White | NA — Not collected
  More than one race | NA — Not collected
  Unknown or Not Reported | NA — Not collected
Region of Enrollment [Number; unit: participants]
  United States | 521

OUTCOME MEASURES:

1. Primary Outcome: High Risk Fall Rate
Description: To determine if the fall rate (as measured by falls per 1000 patient days) for patients designated "high fall risk" decreases with the use of the intervention (Patient is UP fall prevention technology [PUP™ ]) when compared to historical NDNQI data for the prior 12 months ("Benchmark Data") from nursing units where the intervention is being undertaken.
Time Frame: hospital stay (on average 5 days)
Measure: Number; unit: falls/1000 patient days
Arm/Group | Palarum Fall Prevention System
Number analyzed (Participants) | 521
falls/1000 patient days | 0

ADVERSE EVENTS:
Time Frame: There were no adverse events- data was assessed for each individual during their length of stay (avg = 5.4 days)
Description: This was a low risk study- there were no adverse events or mortality related to this study
Arm/Group | Palarum Fall Prevention System
All-Cause Mortality (participants affected / at risk) | 0/521
Serious Adverse Events (participants affected / at risk) | 0/521
Other Adverse Events (participants affected / at risk) | 0/521

LIMITATIONS AND CAVEATS:
Reduced sample size due to having to end study early related to Covid. Sample population is those that agreed to participating in study and those patients admitted to a neuro service line.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03678402/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03678402/SAP_003.pdf